CLINICAL TRIAL: NCT01309555
Title: Easypod Connect: An Australian Multi-centre, Observational Registry to Study Adherence and Long Term Outcomes of Therapy in Paediatric Subjects Using Easypod™ Electromechanical Device for Growth Hormone Treatment
Brief Title: To Assess the Level of Adherence of Subjects Receiving SAIZEN® Via Easypod™ in Australia
Acronym: ECOS AUS
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200104-521
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Growth Disorders
Keywords: Growth disorders; Saizen; easypod™; Growth hormone; Pediatric subject
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: easypod™ — Saizen (Somatropin) as per Summary of Product Characteristics administered by easypod™
  Other Names: Somatropin

SUMMARY:
This is an Australian, Multicentre, Observational Registry to study Adherence and Long Term Outcomes of Therapy in paediatric subjects using easypod™ electromechanical device for growth hormone treatment to assess the level of adherence of subject receiving SAIZEN® via easypod™.

DETAILED DESCRIPTION:
Subjects will be enrolled in a multicenter longitudinal observational registry. Parents/subjects will provide their Informed Consent/assent to upload their data for populationbased analyses and optionally to adhere to a patient adherence support program designed to improve their adherence and, ultimately, clinical outcomes. Adherence data will be primarily derived from the easypod™ device combined with physician data entry of outcome measures. Data will be collected retrospectively and prospectively. This will allow the establishment of adherence profiles and explore the hypothesis that patient adherence support programs improve adherence and subsequent clinical outcomes. Collected data will be also analyzed in a multinational pooled analysis of comparable national studies.

Primary Objective:

• To assess the level of adherence of subjects receiving SAIZEN® via easypod™

Secondary Objectives:

* To describe the impact of adherence on clinical outcomes for subject receiving SAIZEN® via easypod™
* To identify adherence subject profiling based on age, gender, self injection or not, time on treatment, medical history at time of enrollment
* To assess the impact of adherence on Insulin-like Growth Factor 1 (IGF1) (above, below or within normal ranges)

ELIGIBILITY:
Inclusion Criteria:

* Administered growth hormone via the easypod™ electromechanical device according to the SAIZEN® Product Information
* Aged between 2 and 18 years
* Appropriate Informed Consent/Assent provided

Exclusion Criteria:

* Subjects with mature bone age taking growth hormone (i.e. for taking growth hormone for its metabolic effects)
* Contra-indications to SAIZEN® as defined in SAIZEN® Product Information
* Use of an investigational drug or participation in another interventional clinical trial

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric subjects (aged 2-18) who are taking SAIZEN® for registered indications using the Easypod™ electromechanical device.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Mean percent of adherence by subject | At least 6 months and up to 5 years

SECONDARY OUTCOMES:
Correlation of adherence and growth outcome after each year of SAIZEN® treatment with easypod™ | At least 6 months and up to 5 years
  Correlation of adherence and growth outcome (height velocity (HV), height velocity-standard deviation score (HV-SDS), height, change in height (height SDS) after each year of SAIZEN® treatment with easypod™
Subject adherence profile based on age, gender, indication, self-injection or not, time on treatment with easypod™ | At least 6 months and up to 5 years
Correlation of adherence with current IGF-I status (i.e. above, below or within normal ranges) | At least 6 months and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Australia Pty Ltd
Locations (1):
- For Recruiting Locations in Australia, Please Contact the Merck KGaA Communication Center, Australia

REFERENCES:
- [Result] Koledova, E. et al. (2017) Analysis of results from the global, 5-year Easypod™ Connect Observational Study (ECOS) study in children with growth disorders. 10th International Meeting for Pediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Result] Wit, JM. et al. (2017) Effect of adherence on the 2-year growth response to growth hormone treatment in prepubertal children with idiopathic isolated growth hormone deficiency participating in the EasypodTM Connect Observational Study (ECOS). 10th International Meeting of Paediatric Endocrinology; 2017 Sep 14-17; Washington, DC.